CLINICAL TRIAL: NCT06816433
Title: A Phase 2, Multi-center, Multi-arm, Randomized, Placebo-controlled, Double-blind, Adaptive Platform Study to Evaluate the Safety, Tolerability, and Efficacy of Potential Pharmacotherapeutic Interventions in Active-Duty Service Members and Veterans With PTSD
Brief Title: Department of Defense PTSD Adaptive Platform Trial - Intervention D - SLS-002
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Global Coalition for Adaptive Research (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); PPD Development, LP (Industry); Berry Consultants (Other); Idorsia Pharmaceuticals Ltd. (Industry); Cambridge Cognition Ltd (Industry); Citeline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-21-02 (SLS-002)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: SLS-002 is one of multiple interventions that will be tested in this adaptive platform trial (NCT05422612).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The overall 2-stage randomization scheme will be implemented by an unblinded statistician who is otherwise uninvolved in study operations. Participants will be assigned a study number at Screening (Subject ID). In the first stage of randomization, eligible participants who complete screening will be randomly assigned to an open platform cohort for which they are eligible (both site PIs and participants are aware of the cohort assignment) and, within that cohort, the second stage of randomization is to intervention vs placebo (double-blind) using Interactive Response Technology (IRT).
  For this Adaptive Platform Trial (APT), participants assignment to a cohort will not be blinded. The devices used in this cohort may not be visually similar between cohorts and blinding to cohort assignment is not necessary to avoid bias. However, within each cohort, participants, site personnel, contract research personnel and the sponsor will be blind to treatment assignment (intervention vs. placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention D: SLS-002 (Experimental)
  Interventions: Drug: Intervention D SLS-002
- Intervention D: Placebo (Placebo Comparator)
  Interventions: Drug: Intervention D Placebo

INTERVENTIONS:
Drug: Intervention D SLS-002 — SLS-002 will be administered via intranasal administration (one spray per nostril, per device) at 78 mg two times per week for the first eight weeks and then once a week for the last four weeks.
  Other Names: Ketamine
  Arms: Intervention D: SLS-002
Drug: Intervention D Placebo — A matching placebo will be administered via intranasal administration (one spray per nostril, per device) two times per week for the first eight weeks and then once a week for the last four weeks.
  Arms: Intervention D: Placebo

SUMMARY:
This is a Phase 2 randomized, double-blinded, placebo-controlled study that will evaluate multiple potential pharmacotherapeutic interventions for Post Traumatic Stress Disorder (PTSD) utilizing an adaptive platform trial (APT) design.

Intervention D - SLS-002 will assess the safety and efficacy of SLS-002 in participants with PTSD.

Please see NCT05422612 for information on the S-21-02 Master Protocol.

DETAILED DESCRIPTION:
The general structure of this Adaptive Platform Trial (APT) consists of a 30-day Screening Period, a 12-week Platform Treatment Period, and a 4-week Safety Follow-up. The S-21-02 Platform Trial will evaluate the safety and efficacy of multiple investigational products for the treatment of PTSD (see NCT05422612 for Master Protocol information). Participants are randomized among the multiple cohorts in the study and the resulting randomization enables sharing/pooling of control subjects, where all interventions may be compared to a common control (placebo). This record only includes information relevant to the SLS-002 cohort.

Once a participant meets all eligibility criteria for the Master Protocol, eligibility for each currently enrolling intervention cohort is assessed. Eligible participants will be randomized with equal probability into a cohort. Participants randomized to the SLS-002 cohort are then randomly assigned to receive either SLS-002 or placebo (in a ratio of 5:3; intervention:placebo), for the duration of the 12-week treatment period.

Parties interested in having their intervention considered for testing within the Military and Veterans PTSD Adaptive Platform Clinical Trial (M-PACT) should complete a request for information form using this webpage https://citeline.qualtrics.com/jfe/form/SV_8eTQKw6TNug4z42.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria are in addition to the exclusion criteria specified in the Master Protocol (NCT05422612).

1. Is able to complete intranasal administration of study intervention.
2. Is able to refrain from alcohol or cannabis consumption/use on dosing days.
3. Is willing and able to attend dosing visits as outlined in the protocol (twice a week for the first 8 week and then once a week for Weeks 9 through 12) and agrees not to drive a car or operate machinery for 24 hours after receiving the study intervention.

Exclusion Criteria:

The following exclusion criteria are in addition to the exclusion criteria specified in the Master Protocol (NCT05422612).

1. Has a history of seizures (other than childhood febrile seizures).
2. Has a body mass index >40 or <18 kg/m2 at Screening.
3. Has known, uncontrolled hypertension or blood pressure that, in the investigator's judgment, should exclude the subject at Screening or Baseline (blood pressure may be repeated as per the site's standard operating procedures).
4. Has a known history or current finding of cardiovascular disease, cerebrovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, congenital heart disease, ischemic heart disease, cardiac insufficiency, supraventricular, ventricular heart rhythm disorder, prolonged QT syndrome (ie, QTcF >450 msec for males and >470 msec for females) or associated risk factors (ie, hypokalemia, family history of long QT syndrome), syncope, cardiac conduction problems (eg, clinically significant heart block), exercise-related cardiac events including syncope and pre-syncope, clinically significant bradycardia, or other serious cardiac problems.
5. Has a concurrent chronic or acute illness, or other condition (eg, narcolepsy, uncontrolled hyper- or hypothyroidism) that might confound the results of safety assessments conducted in the study.
6. Has any medical condition that could interfere with the absorption of intranasal ketamine (eg, nasal polyps, clinically significant deviated septum [corrected or persistent], or other physical abnormalities of the nose).
7. Has a history of interstitial or ulcerative cystitis, overactive bladder, painful bladder
8. syndrome, chronic pelvic pain, frequent recurrent urinary tract infections, autoimmune disease, active urinary tract infection, history of prostate cancer, bladder cancer or bladder

   a. surgery, or symptoms suggestive of these disorders (eg, high urinary frequency, persistent urge to urinate).
9. Has any history of using ketamine or esketamine. Note previous use of ketamine for anesthesia is allowed.
10. Has known or suspected intolerance or hypersensitivity to the study intervention(s), closely related compounds, or any ingredients.
11. Does not meet or is not willing to comply with the requirements listed in protocol related to prohibited and restricted medications and therapies, as well as required washout periods prior to participation. Prohibited medications and therapies include, but are not limited to, monoamine oxidase inhibitors (MAOIs), chronic/frequent use of opioids or drugs with activity at the opioid receptor, psychostimulants, mood stabilizers/anticonvulsants, antipsychotics, or any medication/therapy that might confound the results of safety assessments conducted in the study. Subjects who have received any of these prohibited medications within 30 days of Screening are excluded from the study. Potent CYP 3A4 inhibitors, including nefazodone and fluvoxamine, are not permitted within 1 week of first dose and until at least 1 day after the last dose. Potent CYP 3A4 inducers, including a. St. John's wort, are not permitted within 30 days of first dose and until at least 1 day after the last dose.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who have undergone or plans to undergo gender reassignment surgery are not eligible.
  Participants who are currently undergoing stable hormone replacement therapy are eligible for inclusion in the study.
Enrollment: 200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Absolute change in the Clinician-Administered PTSD Scale-5-Revised (CAPS-5-R) Past Month total score at Week 12 (Final/Early termination Visit). | 12 Weeks
  A change in PTSD symptom severity from baseline as measured by CAPS-5-R Past Month. The range of the scale is 0-200. The higher the score at baseline, the worse the PTSD severity. The larger the decrease in score from baseline, the better the outcome.
Incidence of new or worsening suicidal thoughts or behaviors as measured by change in Columbia Suicide Severity Rating Scale (C-SSRS) score from baseline. | 12 Weeks
  The C-SSRS is an assessment of suicidal ideation and behavior in clinical and research settings. The C-SSRS consists of 16 questions that ask about suicidal ideation and behaviors (the first 10 questions comprise the ideation subscale and the last 6 comprise the behavior subscale). This 5-item subscale ranges from a minimum of 0 (corresponding to no suicidal ideation) to a maximum of 5 (representing active suicidal ideation with plan and intent).

SECONDARY OUTCOMES:
Frequency of treatment-emergent adverse events (TEAEs). | 12 Weeks
  The TEAEs recorded during the study will be summarized by system organ class, preferred term, and treatment group. Adverse events and medical history will be coded using the most current version of MedDRA.
Severity of treatment-emergent adverse events (TEAEs). | 12 Weeks
  The TEAEs recorded during the study will be summarized by system organ class, preferred term, and treatment group. Adverse events and medical history will be coded using the most current version of MedDRA.
Frequency of serious adverse events (SAEs) | 12 Weeks
  The SAEs recorded during the study will be summarized by system organ class, preferred term, and treatment group. Adverse events and medical history will be coded using the most current version of MedDRA
Severity of serious adverse events (SAEs). | 12 Weeks
  The SAEs recorded during the study will be summarized by system organ class, preferred term, and treatment group. Adverse events and medical history will be coded using the most current version of MedDRA
Relative change from Baseline to Week 12 in CAPS-5-R, Past Month total score. | 12 Weeks
  A relative change in PTSD symptom severity from baseline as measured by the Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R) Past Month. The range of the scale is 0-200. The higher the score at baseline, the worse the PTSD severity. The larger the decrease in score from baseline, the better the outcome.
Number of participants with a Response Rate ≥30% | 12 Weeks
  ≥30% reduction from Baseline to 12 Weeks in the Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R), Past Month total score. The range of the scale is 0-200. The higher the score, the worse the PTSD severity. The larger the decrease in score from baseline, the better the outcome.
Number of participants with a Response Rate ≥50% | 12 Weeks
  ≥50% reduction from Baseline to 12 Weeks in the Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R), Past Month total score. The range of the scale is 0-200. The higher the score, the worse the PTSD severity. The larger the decrease in score from baseline, the better the outcome.
Number of participants Achieving Remission. | 12 Weeks
  Achieving remission: defined as the Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R), Past Month total score <18. The range of the scale is 0-200. The higher the score, the worse the PTSD severity.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Phoenix VA Healthcare System, Phoenix, Arizona
  - Homestead Associates in Research, Inc., Miami, Florida
  - Advanced Discovery Research, Atlanta, Georgia
  - Tripler Army Medical Center (TAMC), Tripler AMC, Hawaii
  - Cincinnati Veteran's Affairs Medical Center, Fort Thomas, Kentucky
  - Walter Reed National Military Medical Center (WRNMC), Bethesda, Maryland
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Wilford Hall Ambulatory Surgical Center (WHASC), San Antonio, Texas
  - Alexander T. Augusta Military Medical Center (ATAMMC):, Fort Belvoir, Virginia
  - Madigan Army Medical Center, Joint Base Lewis McChord, Washington

REFERENCES:
- [Background] Viele K. Allocation in platform trials to maintain comparability across time and eligibility. Stat Med. 2023 Jul 20;42(16):2811-2818. doi: 10.1002/sim.9750. Epub 2023 Apr 23. PMID 37088912